CLINICAL TRIAL: NCT04846959
Title: Risankizumab Pregnancy Exposure Registry: a Prospective Observational Study on the Safety of Risankizumab Exposure in Pregnant Women and Their Offspring
Brief Title: Study to Evaluate Pregnancy Outcomes in Risankizumab Exposed Pregnancies Relative to Those Non-risankizumab Exposed Pregnancies in Women With FDA Approved Indications
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-036
Record Dates: First submitted 2021-04-14; First posted 2021-04-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Plaque Psoriasis, Psoriatic Arthritis, Crohn's Disease, or Other Conditions for Which Risankizumab is an FDA-approved Treatment
Keywords: Pregnancy; Risankizumab; SKYRIZI™; risankizumab-rzaa
MeSH Terms: conditions — Arthritis, Psoriatic; Crohn Disease | interventions — risankizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Pregnant Women Exposed to Risankizumab: Pregnant women of any age in the United States (US) who are diagnosed with plaque psoriasis, psoriatic arthritis, Crohn's disease, or other conditions for which risankizumab is an FDA-approved treatment and exposed to risankizumab at any time during pregnancy.
  Interventions: Drug: Risankizumab
- Pregnant Women Not Exposed to Risankizumab: Pregnant women of any age in the US who are diagnosed with plaque psoriasis, psoriatic arthritis, Crohn's disease, or other conditions for which risankizumab is an FDA-approved treatment and not exposed to risankizumab, but who are exposed to other medications in the same class or line of therapy as risankizumab at any time during pregnancy.
  Interventions: Drug: Comparator

INTERVENTIONS:
Drug: Risankizumab — Subcutaneous Injection
  Other Names: Skyrizi
  Groups: Pregnant Women Exposed to Risankizumab
Drug: Comparator — Subcutaneous or Intravenous Injection
  Groups: Pregnant Women Not Exposed to Risankizumab

SUMMARY:
The objective of this registry is to compare outcomes of risankizumab-exposed pregnancies with those of pregnancies that were not exposed to risankizumab among women with plaque psoriasis, psoriatic arthritis (PsA), Crohn's disease (CD), or other conditions for which risankizumab is an FDA-approved treatment. The registry is designed to estimate the association between risankizumab and maternal, fetal, and infant outcomes by comparing the prevalence rates of these outcomes in the exposed and unexposed populations.

Approximately 818 female participants with pregnancy will be enrolled (409 participants exposed to risankizumab and 409 without exposure) at multiple sites across the United States.

Participants will not receive risankizumab as part of this study. Maternal and fetal outcomes during pregnancy for female participants who received risankizumab or other treatment will be followed for and up to 1 year after delivery

There may be a higher burden for participants in this study compared to standard of care. Participants will attend visits determined by HCPs during the study at a hospital or clinic. The pregnancy outcomes including side effects will be collected during routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

Risankizumab-Exposed Cohort

* US resident.
* Current pregnancy.
* Diagnosis of plaque psoriasis, PsA, CD, or other condition(s) for which Risankizumab is an FDA-approved treatment while the study is recruiting.
* Exposure to risankizumab at any time during pregnancy (at least 1 dose during pregnancy or within 20 weeks prior to conception).

Diseased Comparison Cohort

* US resident.
* Current pregnancy.
* Diagnosis of plaque psoriasis, PsA, CD, or other condition(s) for which Risankizumab is an FDA-approved treatment while the study is recruiting.
* Exposure to other medications in the same class or line of therapy as risankizumab (TNF inhibitors, IL-17 inhibitors, IL-12/23 inhibitor, and other IL-23 inhibitors) at any time during pregnancy (at least 1 dose during pregnancy or prior to pregnancy within a specified time period based on the product's half-life).

Exclusion Criteria:

Risankizumab-Exposed Cohort

* Exposure to other medications in the same class or line of therapy as risankizumab (TNF inhibitors, IL-17 inhibitors, IL-12/23 inhibitor, and other IL-23 inhibitors) at any time during pregnancy (at least 1 dose during pregnancy or prior to pregnancy within a specified time period based on the product's half-life).
* Occurrence of pregnancy outcome prior to enrollment in the registry

Diseased Comparison Cohort

* Exposure to risankizumab at any time during pregnancy (at least 1 dose during pregnancy or within 20 weeks prior to conception).
* Occurrence of pregnancy outcome prior to enrollment in the registry

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise 2 cohorts of pregnant women.
  * One cohort will include pregnant women of any age in the US who are diagnosed with plaque psoriasis, psoriatic arthritis, Crohn's disease, or other conditions for which risankizumab is an FDA-approved treatment and exposed to risankizumab at any time during pregnancy .
  * The second cohort will include pregnant women of any age in the US who are diagnosed with plaque psoriasis, psoriatic arthritis, Crohn's disease, or other conditions for which risankizumab is an FDA-approved treatment and not exposed to risankizumab but who are exposed to other medications in the same class or line of therapy as risankizumab at any time during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 818 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2032-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Major Congenital Malformation (MCM) | Up to 9 months
  MCM is an abnormality of body structure or function that is present at birth, is of prenatal origin (i.e., birth defect), has significant medical, social, or cosmetic consequences for the affected individual, and typically requires medical intervention.

SECONDARY OUTCOMES:
Number of Participants with Minor Congenital Malformation | Up to approximately 2 years (1 year post delivery)
  Minor Congenital Malformation is an anomaly or abnormality of body structure that is present at birth, is of prenatal origin (i.e., birth defect), poses no significant health problem in the neonatal period, and tends to have limited social or cosmetic consequences for the affected individual.
Number of Participants with Stillbirth | Up to 9 months
  Stillbirth is defined by the American College of Obstetricians and Gynecologists (ACOG), an involuntary fetal loss occurring at 20 gestational weeks or greater (>=20 gestational weeks), or, if gestational age is unknown, a fetus weighing 350 g or more (>=350 g).
Number of Participants with Spontaneous Abortion (SAB) | Up to 9 months
  Spontaneous abortion is defined as an involuntary fetal loss or expulsion of products of conception occurring at less than 20 gestational weeks.
Number of Participants with Elective Termination of Pregnancy | Up to 9 months
  Elective termination of pregnancy is defined as an voluntary fetal loss or interruption of pregnancy, including pregnancy termination that occurs electively.
Number of Participants with Preterm Birth | Up to 9 months
  Preterm birth is defined as live birth occurring at less than 37 gestational weeks.
Number of Participants who are Small for Gestational Age (SGA) | Up to 9 months
  SGA is defined as Birth weight less than the 10th percentile for sex and gestational age using standard growth charts for full and preterm live-born infants.
Number of Participants with Neonatal Death | Up to approximately 10 months (one month post delivery)
  Neonatal death is defined as death of a live-born infant within 28 days of life.
Number of Participants with Serious Infection in the First 6 Months of Life | Up to approximately 2 years (1 year post delivery)
  Serious infection is defined as an infection that occurs within an infant's first 6 months of life and results in significant disability, incapacity, or death, is life-threatening, requires inpatient or prolonged hospitalization, or is considered medically important.
Number of Participants with Postnatal Growth Deficiency | Up to approximately 2 years (1 year post-delivery)
  Postnatal growth deficiency is defined as postnatal infant weight less than the 10th percentile for sex and chronological age using standard growth charts.
Number of Participants with Infant Developmental Delay | Up to approximately 2 years (1 year post delivery)
  Infant developmental delay is defined as failure to achieve the developmental milestones for chronological age, as defined by the Center for Disease Control and Prevention (CDC) .

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- United States (2):
  - Evidera, a PPD Business Unit /ID# 238688, Morrisville, North Carolina
  - PPD Development, LP /ID# 232134, Wilmington, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.glowpregnancyregistry.com